CLINICAL TRIAL: NCT04650932
Title: Dual Frequency, Dual Region Deep Brain Stimulation of the Subthalamic Nucleus in Parkinson's Disease
Brief Title: Dual Frequency Stimulation in Parkinson's Disease
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Davis (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1633883
Record Dates: First submitted 2020-11-16; First posted 2020-12-03 (Actual); Last update posted 2025-03-27 (Actual); Status verified 2025-03

CONDITIONS: Parkinson Disease
Keywords: DBS; Deep Brain Stimulation; STN; Subthalamic Nucleus; Parkinson disease; Dual frequency; Dual region; DFDR
MeSH Terms: conditions — Parkinson Disease | interventions — Deep Brain Stimulation

STUDY DESIGN:
Masking Description: Open-label
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Sustained Dual Frequency, Dual Region, Stimulation (Experimental)
  Interventions: Device: Deep brain stimulation

INTERVENTIONS:
Device: Deep brain stimulation — Patients with idiopathic Parkinson's disease who have previously been implanted with the Boston Scientific VerciseTM DBS system for at least 3 months. These patients will already be receiving high-frequency dorsal STN stimulation as part of the standard of care for PD. Once patients have provided consent and are enrolled in this study, they will receive simultaneous low-frequency stimulation of the ventral STN to examine if there are any effects on cognitive performance.
  Other Names: Boston Scientific Vercise DBS

SUMMARY:
Deep brain stimulation (DBS) in the dorsal region of the subthalamic nucleus (STN) is very effective for reducing motor symptoms of Parkinson's disease (PD). Modeling studies suggest that this therapy may result in current spread into the ventral STN, causing altered cognitive processes. As a result, current stimulation parameters often lead to worsening in verbal fluency, executive function, and, particularly, cognitive control. There is evidence suggesting that low frequency oscillatory activity occurs across brain circuits important in integrating information for cognition. Preclinical studies and human recording studies indicate these low frequency theta oscillations drive cognitive control during cognitive tasks. Thus, the purpose of this study is to determine the safety, tolerability, and efficacy of low frequency stimulation (LFS) of the ventral STN alongside standard high frequency stimulation (HFS) of the dorsal STN in patients with PD.

ELIGIBILITY:
Inclusion Criteria:

* Individuals who are 18 years and older
* Individuals with idiopathic Parkinson's Disease who previously underwent implantation with the Boston Scientific VerciseTM DBS system
* Individuals who have been implanted with the Boston Scientific VerciseTM DBS system for at least 3 months
* Individuals diagnosed with advanced PD who had bilateral dorsal subthalamic nucleus DBS surgery, as standard of care for motor improvement, with distal contacts of the electrodes implanted into the ventral STN

Exclusion Criteria:

* Individuals unable to provide consent and/or lack capacity to consent
* Individuals diagnosed with any cognitive or physical impairments that would limit their ability to participate in the cognitive testing
* Individuals who score below 15 on the Montreal Cognitive Assessment Test-Blind
* Individuals who score above 20 on the Center for Epidemiologic Studies Depression Scale
* Pregnant women (note: pregnant women are not candidates for DBS surgery), and prisoners
* Non-English speaking individuals. Cognitive tasks will only be conducted in English.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2022-10-22 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Mean Change from Baseline in Depression Scores on the Center for Epidemiologic Studies Depression Scale (CES-D) | Baseline, Week 2, Week 6, Month 3, and Month 6
  The score of the CES-D will be compared across sessions and a score that rises above 20 (out of 60) will be considered positive for the development of depression.
Mean Change from Baseline in Impulsiveness Scores on the Barratt Impulsiveness Scale (BIS-11) | Baseline, Week 2, Week 6, Month 3, and Month 6
  The score of the BIS-11 will be evaluated across sessions and elevated scores indicate greater impulsivity and risk-taking behavior. The scale involves 30 questions with values from 1-4. Overall scores range from 30-120.
Mean Change from Baseline in Neuropsychiatric Inventory (NPI) | Baseline, Week 2, Week 6, Month 3, and Month 6
  The NPI assesses frequency, change in severity, and distress over 12 neuropsychiatric domains as evaluated by the caregiver. We will look for a significant score reduction in any domain of the NPI.
Mean Change from Baseline in Movement Scores on Part III of the Unified Parkinson's Disease Rating Scale (MDS-UPDRS) | Baseline, Week 2, Week 6, Month 3, and Month 6
  Part III of the MDS-UPDRS consists of 18 areas of motor assessments to assess severity of symptoms. Each score is rated in terms of severity from 0-4, with higher scores indicating higher severity of symptoms. A composite score will be evaluated for changes from baseline.
Mean Change from Baseline in Cognitive Performance Scores on the Montreal Cognitive Assessment - Blind (MoCA) | Baseline, Hour 24, Week 1, Month 1, Month 2, Month 4, and Month 5
  This will be collected via telephone calls. The MoCA-Blind has been validated for telephone administration. We will re-evaluate MoCA-Blind scores during telephone monitoring to assess any changes to cognitive ability. A total score of less than 15 out of a possible 22 indicates greater than mild cognitive impairment.
Mean Change from Baseline in Depression Scores on the CES-D Short Version (CES-D-R10) | Baseline, Hour 24, Week 1, Month 1, Month 2, Month 4, and Month 5
  This will be collected via telephone calls. Patients will be given an unmarked form with questions and will be able to follow along the telephone conversation and answer each question (0-4 severity rating scale) for 10 questions focused on patient affect. A total score greater than 10 (out of 30) indicates the development of depression symptoms.
Mean Change from Baseline in Motor and Non-Motor Aspects of Daily Living Scores on Parts I and II of the MDS-UPDRS | Baseline, Hour 24, Week 1, Month 1, Month 2, Month 4, and Month 5
  This will be collected via telephone calls. Patients will be asked questions relating to motor and non-motor aspects of daily living and to rate the severity of their symptoms on a scale from 0-4, with higher scores indicating higher severity of symptoms. We will assess for changes in the composite score from baseline.

SECONDARY OUTCOMES:
Mean Change from Baseline in Decision-Making Scores on Probabilistic Gambling Task | Baseline, Minute 30, Week 2, Week 6, Month 3, and Month 6
  A patient-specific measure of risk attitude during a gambling task. We will estimate indifference points (win probability at which risky choice is chosen 50% of the time) at each time point and compare to those points during baseline performance on the task.
Mean Change from Baseline in Inter-Temporal Choice Scores on a Temporal Discounting Task | Baseline, Minute 30, Week 2, Week 6, Month 3, and Month 6
  A patient-specific measure of risk attitude during a temporal preferences task. We will examine the area under the curve of the empirical discount functions of 'larger later' rewards and 'smaller sooner' rewards. Smaller values indicate increased preference for smaller sooner over larger later rewards. Scores will be compared to baseline performance on the task.
Mean Change from Baseline in Verbal Fluency Scores on Word Generation Task | Baseline, Minute 30, Week 2, Week 6, Month 3, and Month 6
  The average number of words generated in a 1-minute time frame.

CONTACTS AND LOCATIONS:
Overall Officials: Kiarash Shahlaie, MD, PhD, Principal Investigator — University of California, Davis
Locations (1):
- UC Davis Health, Sacramento, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Scangos KW, Carter CS, Gurkoff G, Zhang L, Shahlaie K. A pilot study of subthalamic theta frequency deep brain stimulation for cognitive dysfunction in Parkinson's disease. Brain Stimul. 2018 Mar-Apr;11(2):456-458. doi: 10.1016/j.brs.2017.11.014. Epub 2017 Nov 23. No abstract available. PMID 29203130
- [Background] Bergman H, Wichmann T, DeLong MR. Reversal of experimental parkinsonism by lesions of the subthalamic nucleus. Science. 1990 Sep 21;249(4975):1436-8. doi: 10.1126/science.2402638.
- [Background] Le Jeune F, Peron J, Grandjean D, Drapier S, Haegelen C, Garin E, Millet B, Verin M. Subthalamic nucleus stimulation affects limbic and associative circuits: a PET study. Eur J Nucl Med Mol Imaging. 2010 Aug;37(8):1512-20. doi: 10.1007/s00259-010-1436-y. Epub 2010 Mar 28. PMID 20349231
- [Background] Sharma AK, Reams RY, Jordan WH, Miller MA, Thacker HL, Snyder PW. Mesial temporal lobe epilepsy: pathogenesis, induced rodent models and lesions. Toxicol Pathol. 2007 Dec;35(7):984-99. doi: 10.1080/01926230701748305. PMID 18098044
- [Background] Volkmann J. Deep brain stimulation for the treatment of Parkinson's disease. J Clin Neurophysiol. 2004 Jan-Feb;21(1):6-17. doi: 10.1097/00004691-200401000-00003. PMID 15097290
- [Background] Frankemolle AM, Wu J, Noecker AM, Voelcker-Rehage C, Ho JC, Vitek JL, McIntyre CC, Alberts JL. Reversing cognitive-motor impairments in Parkinson's disease patients using a computational modelling approach to deep brain stimulation programming. Brain. 2010 Mar;133(Pt 3):746-61. doi: 10.1093/brain/awp315. Epub 2010 Jan 7. PMID 20061324
- [Background] Holz EM, Glennon M, Prendergast K, Sauseng P. Theta-gamma phase synchronization during memory matching in visual working memory. Neuroimage. 2010 Aug 1;52(1):326-35. doi: 10.1016/j.neuroimage.2010.04.003. Epub 2010 Apr 9. PMID 20382239
- [Background] Colgin LL. Mechanisms and functions of theta rhythms. Annu Rev Neurosci. 2013 Jul 8;36:295-312. doi: 10.1146/annurev-neuro-062012-170330. Epub 2013 May 29. PMID 23724998
- [Background] Lee DJ, Gurkoff GG, Izadi A, Seidl SE, Echeverri A, Melnik M, Berman RF, Ekstrom AD, Muizelaar JP, Lyeth BG, Shahlaie K. Septohippocampal Neuromodulation Improves Cognition after Traumatic Brain Injury. J Neurotrauma. 2015 Nov 15;32(22):1822-32. doi: 10.1089/neu.2014.3744. Epub 2015 Sep 2. PMID 26096267
- [Background] Izadi A, Pevzner A, Lee DJ, Ekstrom AD, Shahlaie K, Gurkoff GG. Medial septal stimulation increases seizure threshold and improves cognition in epileptic rats. Brain Stimul. 2019 May-Jun;12(3):735-742. doi: 10.1016/j.brs.2019.01.005. Epub 2019 Jan 17. PMID 30733144
- [Background] Cohen MX, Cavanagh JF. Single-trial regression elucidates the role of prefrontal theta oscillations in response conflict. Front Psychol. 2011 Feb 28;2:30. doi: 10.3389/fpsyg.2011.00030. eCollection 2011. PMID 21713190
- [Background] Zavala BA, Tan H, Little S, Ashkan K, Hariz M, Foltynie T, Zrinzo L, Zaghloul KA, Brown P. Midline frontal cortex low-frequency activity drives subthalamic nucleus oscillations during conflict. J Neurosci. 2014 May 21;34(21):7322-33. doi: 10.1523/JNEUROSCI.1169-14.2014. PMID 24849364
- [Background] Zavala B, Brittain JS, Jenkinson N, Ashkan K, Foltynie T, Limousin P, Zrinzo L, Green AL, Aziz T, Zaghloul K, Brown P. Subthalamic nucleus local field potential activity during the Eriksen flanker task reveals a novel role for theta phase during conflict monitoring. J Neurosci. 2013 Sep 11;33(37):14758-66. doi: 10.1523/JNEUROSCI.1036-13.2013. PMID 24027276
- [Background] Frank MJ, Samanta J, Moustafa AA, Sherman SJ. Hold your horses: impulsivity, deep brain stimulation, and medication in parkinsonism. Science. 2007 Nov 23;318(5854):1309-12. doi: 10.1126/science.1146157. Epub 2007 Oct 25. PMID 17962524
- [Background] Smarr KL, Keefer AL. Measures of depression and depressive symptoms: Beck Depression Inventory-II (BDI-II), Center for Epidemiologic Studies Depression Scale (CES-D), Geriatric Depression Scale (GDS), Hospital Anxiety and Depression Scale (HADS), and Patient Health Questionnaire-9 (PHQ-9). Arthritis Care Res (Hoboken). 2011 Nov;63 Suppl 11:S454-66. doi: 10.1002/acr.20556. No abstract available. PMID 22588766
- [Background] Miller WC, Anton HA, Townson AF. Measurement properties of the CESD scale among individuals with spinal cord injury. Spinal Cord. 2008 Apr;46(4):287-92. doi: 10.1038/sj.sc.3102127. Epub 2007 Oct 2. PMID 17909558
- [Background] Bjorgvinsson T, Kertz SJ, Bigda-Peyton JS, McCoy KL, Aderka IM. Psychometric properties of the CES-D-10 in a psychiatric sample. Assessment. 2013 Aug;20(4):429-36. doi: 10.1177/1073191113481998. Epub 2013 Mar 18. PMID 23513010
- [Background] Pendlebury ST, Welch SJ, Cuthbertson FC, Mariz J, Mehta Z, Rothwell PM. Telephone assessment of cognition after transient ischemic attack and stroke: modified telephone interview of cognitive status and telephone Montreal Cognitive Assessment versus face-to-face Montreal Cognitive Assessment and neuropsychological battery. Stroke. 2013 Jan;44(1):227-9. doi: 10.1161/STROKEAHA.112.673384. Epub 2012 Nov 8. PMID 23138443
- [Background] Pote I, Torkamani M, Kefalopoulou ZM, Zrinzo L, Limousin-Dowsey P, Foltynie T, Speekenbrink M, Jahanshahi M. Subthalamic nucleus deep brain stimulation induces impulsive action when patients with Parkinson's disease act under speed pressure. Exp Brain Res. 2016 Jul;234(7):1837-1848. doi: 10.1007/s00221-016-4577-9. Epub 2016 Feb 18. PMID 26892884
- [Background] Peters J, D'Esposito M. Effects of Medial Orbitofrontal Cortex Lesions on Self-Control in Intertemporal Choice. Curr Biol. 2016 Oct 10;26(19):2625-2628. doi: 10.1016/j.cub.2016.07.035. Epub 2016 Sep 1. PMID 27593380
- [Background] Seymour B, Barbe M, Dayan P, Shiner T, Dolan R, Fink GR. Deep brain stimulation of the subthalamic nucleus modulates sensitivity to decision outcome value in Parkinson's disease. Sci Rep. 2016 Sep 14;6:32509. doi: 10.1038/srep32509. PMID 27624437
- [Background] Ehlen F, Schoenecker T, Kuhn AA, Klostermann F. Differential effects of deep brain stimulation on verbal fluency. Brain Lang. 2014 Jul;134:23-33. doi: 10.1016/j.bandl.2014.04.002. Epub 2014 May 9. PMID 24815947
- [Background] Laxton AW, Lozano AM. Deep brain stimulation for the treatment of Alzheimer disease and dementias. World Neurosurg. 2013 Sep-Oct;80(3-4):S28.e1-8. doi: 10.1016/j.wneu.2012.06.028. Epub 2012 Jun 19. PMID 22722036
- [Background] Temperli P, Ghika J, Villemure JG, Burkhard PR, Bogousslavsky J, Vingerhoets FJ. How do parkinsonian signs return after discontinuation of subthalamic DBS? Neurology. 2003 Jan 14;60(1):78-81. doi: 10.1212/wnl.60.1.78. PMID 12525722
- [Background] Smeding HM, Speelman JD, Koning-Haanstra M, Schuurman PR, Nijssen P, van Laar T, Schmand B. Neuropsychological effects of bilateral STN stimulation in Parkinson disease: a controlled study. Neurology. 2006 Jun 27;66(12):1830-6. doi: 10.1212/01.wnl.0000234881.77830.66. PMID 16801645
- [Background] Strutt AM, Simpson R, Jankovic J, York MK. Changes in cognitive-emotional and physiological symptoms of depression following STN-DBS for the treatment of Parkinson's disease. Eur J Neurol. 2012 Jan;19(1):121-7. doi: 10.1111/j.1468-1331.2011.03447.x. Epub 2011 Jun 11. PMID 21668586